CLINICAL TRIAL: NCT05575427
Title: Efficacy of Combination Therapy With Minocycline for Treatment of Stenotrophomonas Maltophilia Infections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SI-CEU-01-2022
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Hospital Infections
Keywords: Minocycline; Stenotrophomonas maltophilia
MeSH Terms: conditions — Cross Infection; cyclopia sequence | interventions — Minocycline; Levofloxacin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: A Phase 4 Randomized, Double blind, Placebo Controlled
Who Masked: Participant, Investigator
Masking Description: Double blind, Placebo Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination therapy with minocycline (Experimental): Minocycline oral 50 mg per capsule
  4 capsules oral stat then 2 capsules oral every 12 hours
  duration 7-28 days
  Interventions: Drug: Minocycline; Drug: Levofloxacin or Cotrimoxazole
- Monotherapy plus placebo (Active Comparator): Patients were treated Stenotrophomonas maltophilia infection with standard monotherapy either levofloxacin or Trimethoprim/sulfamethoxazole plus placebo
  Interventions: Drug: Levofloxacin or Cotrimoxazole; Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — The patients will receive minocycline oral between 7-28 days
  Other Names: Mino
  Arms: Combination therapy with minocycline
Drug: Levofloxacin or Cotrimoxazole — The patients will receive levofloxacin or cotrimoxazole oral between 7-28 days
  Other Names: Cravit or Bactrim
Drug: Placebo — Capsule without active compound
  Arms: Monotherapy plus placebo

SUMMARY:
The objective of the study is to evaluate the efficacy of minocycline for treatment Stenotrophomonas maltophilia infection. The hypothesis of study is the combination therapy with minocycline would be better than the monotherapy for treatment Stenotrophomonas maltophilia infection.

DETAILED DESCRIPTION:
* Investigator inform patient or their relatives about all topics in project, eligible criteria, method, material and monitoring treatment.
* After patient or their relatives are appreciated to join this project, patients will be randomly allocated to either levofloxacin or cotrimoxazole plus placebo (monotherapy plus placebo) or levofloxacin or cotrimoxazole plus minocycline (combination therapy).
* Duration of treatment is determined by site and severity of infection, approximately 7-28 days.
* Sample size calculation, by two independent proportions formula, the investigators estimate the mortality rate about 54 % in monotherapy group and mortality rate about 27 % in combination therapy with minocycline group, with 2-sided 95% Confidence interval; therefore,51 persons are needed each group.
* The investigators estimate gather data about 112 persons. (56 participants with monotherapy and 56 participants with combination therapy (minocycline plus another antibiotic drug from intervention trial))
* The categorical variables are reported as frequencies and percentages, while continuous variables are reported as means ± standard deviations for normally distributed data and median ± range for non-normally distributed data. The data collected from patients are compared using Chi-square tests or Fisher's exact tests for categorical variables and using t-tests or Mann-Whitney U-tests for continuous variables.
* During the study is performing, all unexpected adverse event definitely report to Siriraj institutional Review Board immediately, in addition to subjects or their relatives.

ELIGIBILITY:
Inclusion Criteria:

* The infection caused by Stenotrophomonas maltophilia
* The duration of treatment approximately between 7-28 days
* The patients can take minocycline capsule via oral or nasogastric tube feeding.
* The patients are anticipated to live more than 48 hrs after participation.
* In case of an antibiotic drug administration for treatment Stenotrophomonas maltophilia beforehand, it should not exceed 48 hrs.
* All of participants should be willing to join this project.

Exclusion Criteria:

* Pregnancy and lactation
* The patients with active hepatitis
* The patients with history of minocycline allergy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
mortality rate | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  mortality rate of S. maltophilia infected patients receiving treatment at day 28

SECONDARY OUTCOMES:
microbiological clearance | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  we perform culture and staining to assess bacterial clearance after apply the study drug
adverse drug reactions | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  we assess adverse drug reactions in 2 aspects; nephrotoxicity and hepatotoxicity

CONTACTS AND LOCATIONS:
Overall Officials: Adhiratha Boonyasiri, MD, Principal Investigator — Department of research, Faculty of Medicine Siriraj hospital, Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Junco SJ, Bowman MC, Turner RB. Clinical outcomes of Stenotrophomonas maltophilia infection treated with trimethoprim/sulfamethoxazole, minocycline, or fluoroquinolone monotherapy. Int J Antimicrob Agents. 2021 Aug;58(2):106367. doi: 10.1016/j.ijantimicag.2021.106367. Epub 2021 May 28. PMID 34058337
- [Background] Insuwanno W, Kiratisin P, Jitmuang A. Stenotrophomonas maltophilia Infections: Clinical Characteristics and Factors Associated with Mortality of Hospitalized Patients. Infect Drug Resist. 2020 May 28;13:1559-1566. doi: 10.2147/IDR.S253949. eCollection 2020. PMID 32547125